CLINICAL TRIAL: NCT01144468
Title: Effects of Exemestane on Bone Strength in Postmenopausal Women at Increased Risk of Developing Breast Cancer
Brief Title: Effects of Exemestane on Bone Strength
Acronym: MAP3BSS
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Breast Cancer Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: 07-0168
Record Dates: First submitted 2010-06-11; First posted 2010-06-15 (Estimated); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2022-11

CONDITIONS: Osteoporosis; Breast Cancer
Keywords: breast cancer prevention; osteoporosis
MeSH Terms: conditions — Osteoporosis; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MAP3 Participants: study participants in the MAP.3 study are randomly assigned to either placebo or 25 mg exemestane daily for 5 years. Allocation is blinded. We are following 354 of these study participants and are blinded to treatment allocation.

SUMMARY:
The NCIC CTG was conducting an international breast cancer prevention trial (MAP.3) examining the effects of a new therapy (exemestane) for breast cancer prevention in postmenopausal women at increased risk of developing this disease. Results showed that after a median follow up of 35 months, exemestane was superior to placebo in breast cancer prevention. Exemestane blocks estrogen production, which may be beneficial for preventing breast cancer, but may have negative effects on bone. As postmenopausal women are at risk for developing osteoporosis, determining whether exemestane causes bones to weaken is crucial for women considering it for long-term use. Dr. Cheung's team followed the bone health of 354 women in MAP.3 in detail over 2 years and found that volumetric bone mineral density (by high resolution peripheral quantitative computer tomography (HR-pQCT) at the radius and tibia as well as areal bone mineral density by dual energy x-ray absorptiometry (DXA) at the hip and spine decreased significantly with the use of exemestane. The long term effects of exemestane on bone will be examined up to 5 years of therapy and then 2 years post therapy to delineate the effects of exemestane on bone strength. This research will inform us on the safety of exemestane for breast cancer prevention.

DETAILED DESCRIPTION:
Aromatase inhibitors (AIs) substantially decrease estrogen levels in postmenopausal women; thus, they have the potential to prevent breast cancer, but they also have the potential to adversely affect bone. Previous animal data from our group suggests that exemestane, a steroid AI, may have a more favourable effect on bone metabolism than the non-steroidal AIs. Over the past few years, we have been conducting a 2-year companion study in a subset of women participating in the 5-year MAP.3 trial-- a primary breast cancer prevention trial conducted by the NCIC Clinical Trials Group (NCIC CTG) to examine the effects of exemestane on the prevention of breast cancer. This companion study is conducted at 3 geographic locations (Toronto, Canada; Mayo Clinic in Rochester (US) and at the University of California Davis in California (US)) in postmenopausal women who do not have osteoporosis at baseline, to investigate the effects of exemestane on bone structure and density in the first 2 years of taking exemestane.

On November 5 2010, the MAP.3 study reached an early primary breast cancer event-driven endpoint. Data analysis conducted March 2011 showed that after a median follow up of 35 months, exemestane was superior to placebo in breast cancer prevention. Based upon the positive results of the MAP.3 trial, and the relatively low incidence of adverse events seen in women receiving exemestane as compared to those receiving placebo, the trial committee and NCIC CTG have agreed not to close the study. Instead, a modified observational study will continue. We have also extended this 2-year study for another 3 years. Recent data suggests that there is a difference in changes in BMD (and perhaps fractures) in women with breast cancer, with the earlier effects (< 2 years) being worse than the late effects. As exemestane was found to be effective in the prevention of breast cancer, it is likely going to be used for 5 years. By extending this companion study for another 3 years, we will be able to determine the long term (up to 5 years) effects of exemestane on bone structure and density, and to compare the effects observed from 2 to 5 years of follow-up to those observed from baseline to 2 years.

The primary objectives of our original 2-year study and this extension study are to determine whether exemestane will cause a clinically and statistically significant difference in percent change in total volumetric bone mineral density (BMD) at the distal radius as measured by high-resolution peripheral quantitative computed tomography (HRpQCT) from baseline to 2 years and from 2 to 5 years, and 2 years post therapy,as compared to placebo. Our secondary objectives are: 1) to determine the effects of exemestane on cortical and trabecular volumetric BMD as measured by pQCT scans at 1, 2, 3 and 5 years; 2) to examine the effects of exemestane on other bone geometric parameters such as cortical thickness, trabecular thickness, trabecular separation and trabecular number at 1, 2, 3 and 5 years; 3) to investigate the effect of exemestane on the percent change in BMD at the lumbar spine (L1-L4) and the total hip as measured by dual energy X-ray absorptiometry (DXA) from baseline to 1, 2, 3 and 5 years as compared to placebo; and 4) to determine the effect of 2 years of exemestane on bone strength index as compared to placebo. We will also compare the early (baseline to 2 years) and late (2 to 5 years) effects of exemestane on bone. All participants in this companion study are provided with calcium and vitamin D supplementation. Measurements of volumetric BMDs and bone geometric parameters are obtained by HRpQCT using Xtreme CT, and measurements of areal BMDs are obtained by DXA using Hologic or Lunar densitometers at baseline, 1, 2, 3 and 5 years, according to standard protocols.

The results of the proposed extension to the companion study will help us understand the long term effects and long term safety of exemestane on bone health in postmenopausal women at risk of developing breast cancer. Data on healthy postmenopausal women taking long term (2-5 years) exemestane does not exist at this time. Information from this study will help clinicians and women weigh the risks and benefits of using exemestane and make informed decisions regarding breast cancer prevention.

ELIGIBILITY:
Inclusion Criteria:

Women participating in the MAP.3 clinical trial at centres with access to HR-pQCT

Exclusion Criteria:

1. Women with osteoporosis;
2. Women with T-score of -2.0 or below at the lumbar spine (L1-L4), total hip or femoral neck;
3. Women with a fragility fracture after age 40;
4. Women who have been on any bone drug, such as hormone replacement therapy, selective estrogen receptor modulators, bisphosphonates, teriparatide, parathyroid hormone, sodium fluoride, strontium, calcitonin and high dose vitamin D (more than 2000iu of vitamin D3 daily),in the past 3 months;
5. Women who have ever been on a bisphosphonate for more than 6 months;
6. Women who have ever been on strontium for more than 1 month;
7. Women who are on chronic oral steroids (the equivalent of 5mg of prednisone a day or higher for more than 2 weeks within the past 6 months and will likely require ongoing therapy);
8. Women with Paget's disease, Cushing's disease, hyperparathyroidism, uncontrolled hyperthyroidism or other metabolic bone diseases;
9. Women with decompensated diseases of the liver, bowel, kidney, pancreas, lung, or heart.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women randomized to the MAP.3 study from 5 participating locations were consecutively approached for participation in this companion study.
Sampling Method: Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2007-04; Primary Completion 2013-05 (Actual); Study Completion 2022-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela MW Cheung, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (4):
- United States (2):
  - University of California Davis, Sacramento, California
  - Mayo Clinic, Rochester, Minnesota
- Canada (2):
  - University Health Network, TGH, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario

REFERENCES:
- [Background] Goss PE, Ingle JN, Ales-Martinez JE, Cheung AM, Chlebowski RT, Wactawski-Wende J, McTiernan A, Robbins J, Johnson KC, Martin LW, Winquist E, Sarto GE, Garber JE, Fabian CJ, Pujol P, Maunsell E, Farmer P, Gelmon KA, Tu D, Richardson H; NCIC CTG MAP.3 Study Investigators. Exemestane for breast-cancer prevention in postmenopausal women. N Engl J Med. 2011 Jun 23;364(25):2381-91. doi: 10.1056/NEJMoa1103507. Epub 2011 Jun 4. PMID 21639806
- [Result] Cheung AM, Tile L, Cardew S, Pruthi S, Robbins J, Tomlinson G, Kapral MK, Khosla S, Majumdar S, Erlandson M, Scher J, Hu H, Demaras A, Lickley L, Bordeleau L, Elser C, Ingle J, Richardson H, Goss PE. Bone density and structure in healthy postmenopausal women treated with exemestane for the primary prevention of breast cancer: a nested substudy of the MAP.3 randomised controlled trial. Lancet Oncol. 2012 Mar;13(3):275-84. doi: 10.1016/S1470-2045(11)70389-8. Epub 2012 Feb 7. PMID 22318095

RESULTS

PARTICIPANT FLOW:
Groups:
- Exemestane; Placebo: In MAP.3 participants were randomly assigned to 25 mg exemestane daily or placebo for 5 years.
Period: Overall Study
Arm/Group | Exemestane | Placebo
Started | 176 | 175
Completed | 124 | 118
Not Completed | 52 | 57
Not completed — Lost to Follow-up | 4 | 7
Not completed — Adverse Event | 3 | 2
Not completed — did not reach 2 year follow up at time of clinical cut off | 45 | 48

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exemestane 25 mg Daily | Placebo | Total
Number analyzed (Participants) | 176 | 175 | 351
Age, Continuous [Mean (Full Range); unit: years] | 61.3 [59.4 to 65.4] | 61.1 [59.2 to 63.9] | 61.2 [59.2 to 65.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176 | 175 | 351
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 00 | 0 | 0
  White | 166 | 162 | 328
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 13 | 23

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Total Volumetric Bone Mineral Density (BMD) Measured by High Resolution Peripheral Quantitative Computer Tomography (HR-PQCT) From Baseline to 24 Months
Description: Mean percent change in total volumetric bone mineral density (BMD) measured by high resolution peripheral quantitative computer tomography )HR-pQCT from baseline to 24 months
Time Frame: 24 months
Population: This is an observational study of participants in the MAP.3 breast cancer prevention randomized controlled trial.
  In MAP.3 participants were randomly assigned to either placebo or 25 mg exemestane daily for 5 years. Allocation was blinded. We are following 354 of these study participants and are blinded to treatment allocation.
Measure: Mean (95% Confidence Interval); unit: mean percent change
Arm/Group | MAP3 Participants on 25 mg Exemestane Daily | MAP3 Participants on Placebo
Number analyzed (Participants) | 176 | 175
mean percent change | -6.1 [-7.0 to -5.2] | -1.8 [-2.4 to -1.2]

ADVERSE EVENTS:
Time Frame: 2 years
Description: Women discontinued the study if their lumbar spine, total hip, or femoral neck areal BMD dropped 10% or more in the preceding year, their T-scores fell to or below -2·5, or if they sustained fragility fractures or started taking drugs for bone-related disorders
Groups:
- MAP3 Participants on 25 mg Exemestane Daily: MAP3 treatment arm
- MAP3 Participants on Placebo: MAP3 placebo arm
Arm/Group | MAP3 Participants on 25 mg Exemestane Daily | MAP3 Participants on Placebo
All-Cause Mortality (participants affected / at risk) | 0/176 | 0/175
Serious Adverse Events (participants affected / at risk) | 0/176 | 0/175
Other Adverse Events (participants affected / at risk) | 3/176 | 2/175
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MAP3 Participants on 25 mg Exemestane Daily (N=176) | MAP3 Participants on Placebo (N=175)
Bone related adverse event (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No